CLINICAL TRIAL: NCT05311488
Title: Early Detection of Peripheral Neuropathy in Hereditary Transthyretin Amyloidosis
Brief Title: Early Detection of Neuropathy in ATTRv
Acronym: EDONA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 849579
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Amyloidosis, Transthyretin-Related
Keywords: transthryretin; Hereditary transthyretin amyloidosis; TTRv; familial amyloid polyneuropathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloid Neuropathies, Familial | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be processed, and serum will be stored according to PDMDC GeneticsBiobank protocol. The serum will be assayed by ultrasensitive single molecule array (Simoa NF-Light® assay, Quanterix, Lexington, MA) to determine NF-L concentration. Samples will be tested in duplicate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic TTRv: Patients with known TTR mutations and neuropathy
  Interventions: Diagnostic Test: neurofilament light chain; Diagnostic Test: In-vivo Meissner Corpuscle imaging; Diagnostic Test: Nerve conduction study
- Asymptomatic TTRv: Patients with TTR mutation and no symptoms within less than 10 years of typical onset of disease
  Interventions: Diagnostic Test: neurofilament light chain; Diagnostic Test: In-vivo Meissner Corpuscle imaging; Diagnostic Test: Nerve conduction study
- Healthy controls: Age and sex matched healthy controls without neuropathy or other neurological disorder.
  Interventions: Diagnostic Test: neurofilament light chain; Diagnostic Test: In-vivo Meissner Corpuscle imaging; Diagnostic Test: Nerve conduction study

INTERVENTIONS:
Diagnostic Test: neurofilament light chain — Blood test
Diagnostic Test: In-vivo Meissner Corpuscle imaging — Imaging
Diagnostic Test: Nerve conduction study — Nerve conduction study

SUMMARY:
The purpose of the study is to evaluate and compare different tools that are used to detect evidence of peripheral neuropathy in patients with TTRv.

DETAILED DESCRIPTION:
Early detection of peripheral neuropathy in patients with TTRv is important to support initiation of therapy that alters the course of the disease. Current tools used to detect peripheral neuropathy may not be sensitive, especially in very early and distal peripheral neuropathy. This study will compare different methods of assessing for peripheral neuropathy including using in-vivo reflectance confocal microscopy to assess for meissner corpuscles, serum neurofilament light chain, quantitative sensory testing, neuropathy impairement scores, nerve conduction studies and quality of life and symptoms questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Patients with known TTR mutations and neuropathy

1. Patients with TTR mutation and no symptoms within less than 10 years of typical onset of disease
2. Age criteria must meet the following:

   * Non V122I mutations, Age 40 or older.
   * V122 I mutations, 55 or older.

Healthy persons without neuropathy

1. The following distribution of age ranges will be considered when enrolling healthy participants:

   * 5 patients age 30-40
   * 5 patients age 40-50
   * 5 patients age 50-60
   * 5 patients age 60-70
2. Healthy control subjects for this study are defined as subjects with no symptoms of neuropathy or risk factors for neuropathy such as family history of hereditary neuropathy, chemotherapy, diabetes, autoimmune disease, or vitamin deficiency. Their status will be verified by medical records review.

Exclusion Criteria:

1. Patients with neuropathy other than TTR amyloid
2. Subjects with risk factors for neuropathy (diabetes, history of neuropathy in the family, neurotoxic drugs) or with neurological disorder associated with elevated NFL

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ATTRv symptomatic, asymptomatic and control.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2029-02-14 (Estimated)

PRIMARY OUTCOMES:
Change in Serum neurofilament light chain | 12 months
  Change in Serum neurofilament light chain concentration at 12 months
Meissner corpuscles | 12 months
  Change in Meissner corpuscles density at 12 months

SECONDARY OUTCOMES:
Quantitative sensory testing | 12 months
  Testing of vibratory sensation using a tuning fork, testing of light touch using neurofilament
Neuropathy symptoms questionnaire | 12 months
  Questionnaire that assess symptoms of neuropathy and severity.
Neuropathy impairment score | 12 months
  Neurological examination reporting motor strength, reflexes and sensation. Scale ranges from 0 (normal) to 244, with a higher score indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Chafic Karam, MD, Principal Investigator — University of Pennsylvania; Brian Drachman, Principal Investigator — University of Pennsylvania; Sami Khella, MD, Principal Investigator — University of Pennsylvania; Janice Pieretti, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided